CLINICAL TRIAL: NCT07390175
Title: Ablación de la fibrilación Cardiaca Humana Basada en Modelos de organización jerárquica de la excitación Tisular.
Brief Title: Ablation of Human Cardiac Fibrillation Based on Models of Hierarchical Organization of Tissue Excitation
Acronym: TerFib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Instituto de Salud Carlos III, Ministerio de Sanidad, Spanish Goverment. (Unknown)
Responsible Party: Principal Investigator, Daivd Calvo Cuervo, Cardiologist electrophysiologist, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TerFib_Hyerarchy; 80/18 (Other: HUPA)
Record Dates: First submitted 2026-01-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Ablation Treatment; TerFib_Hyerarchy
Keywords: Hierarchical organization of tissue excitation; Atrial Fibrillation (AF); Ablation; TerFib_Hyerarchy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CPVI only) (Active Comparator): Modifications in fibrillation dynamics induced by CPVI will be evaluated. Therefore, an experimental protocol will be carried out in which, once CPVI has been completed, a new acquisition of non-invasive maps will be performed to characterize basal fibrillation dynamics and those under adenosine
  Interventions: Procedure: Control group ablation
- Active group (CPVI plus extrapulmonary ablation of DFASI domains) (Experimental): Modifications in fibrillation dynamics induced by ablation distributed along the points of singularity of the maintaining reentries (or their inclusion in the CPVI if applicable) will be evaluated, as suggested by our preliminary results (Calvo D et al. Sci Rep. 2025 Dec 16;15(1):43892). Therefore, an experimental protocol will be carried out in which each DFASI reentrant domain will be addressed sequentially. After each ablation set, a new evaluation of noninvasive hierarchical organization patterns will be performed by acquiring new CardioInsight maps in AF
  Interventions: Procedure: Active group ablation

INTERVENTIONS:
Procedure: Active group ablation — In patients in the active group, changes in fibrillation dynamics induced by CPVI and ablation of DFASI domains will be evaluated, as suggested by our preliminary results (Calvo D et al. Sci Rep. 2025 Dec 16;15(1):43892). Therefore, an experimental protocol will be carried out in which, after CPVI, each DFASI domain will be addressed sequentially. The following will be determined: a) changes in hierarchical organization levels, b) the formation of new DFASI domains; c) if AF ends after ablation, the termination mechanisms will be described. Once all ablation sets on the identified DFASI reentrant domains have been completed, noninvasive maps will be acquired under the effect of adenosine in order to compare fibrillatory dynamics under basal adenosine vs. post-ablation.
  Arms: Active group (CPVI plus extrapulmonary ablation of DFASI domains)
Procedure: Control group ablation — Therefore, an experimental protocol will be carried out in which, once the CPVI has been completed, a new acquisition of non-invasive maps will be performed to characterize the basal fibrillation dynamics and those under adenosine.
  Arms: Control group (CPVI only)

SUMMARY:
The mechanisms that maintain persistent atrial fibrillation (AF) in humans remain unknown. In the research project PI18/01268 funded in the previous call for Strategic Action in Health, the group has demonstrated that the hierarchical organization of (i) rotational domains, (ii) frequency domains and (iii) physiological responses to pharmacological provocation with adenosine, allow the identification of domains of high-frequency reentrant activity (hereinafter "DFASI domains") maintainers of AF. As a result, the investigators have developed non-invasive technological models and quantitative indices (currently both subject to patent evaluation; United States Patent and Trademark Office, Application number 63/422,563) for the efficient localization of these domains, whose therapeutic approach through ablation has allowed to improve the clinical results of the patients studied, safely without increase in complications (Calvo D et al. Sci Rep. 2025 Dec 16;15(1):43892). Likewise, and in response to the objectives of the PI18/01268 project, the investigators have identified hierarchical organization patterns in human ventricular fibrillation (VF) that indicate the existence of universal fibrillatory mechanisms, opening the door to new therapeutic opportunities (Europace 2022;24[11]:1788-1799).

DETAILED DESCRIPTION:
The present research project proposes to characterize the physiology of persistent human AF after therapeutic interaction (ablation) with the "DFASI domains", exploring its impact on the dynamics and maintenance of AF in patients. The investigators propose to reveal the physiological mechanisms by which this interaction improves the clinical outcomes of our patients (Objective 1), which will allow the development of more efficient ablation strategies (Objective 2). Likewise, preclinical models developed by our group in collaboration with the National Center for Cardiovascular Research support the translation of our technological developments to the field of human VF. Therefore, in the present research project the investigators propose to explore the physiological significance of "DFSI domains" in patients with recurrent VF and the eventual development of efficient ablative therapies (Objective 3). With the proposed objectives, the project addresses the challenges posed in the diagnosis and treatment of cardiovascular diseases within the National Health System, in the context of a prevalent pathology (cardiac fibrillation) with high morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with persistent AF lasting more than 6 months at the time of the experimental protocol (uninterrupted persistent AF) and clinical indication for an AF ablation procedure.

or

-Patients over 18 years of age with recurrent VF/VT and poor control with conventional pharmacological measures.

Exclusion Criteria:

* Lack of patient consent to participate in the study.
* In patients with persistent AF, contraindication for the use of adenosine.
* AF/VF/VPT secondary to endocrine-metabolic disorders and/or severe systemic disease (thyrotoxicosis, sepsis, pulmonary thromboembolism, etc.).
* Contraindications for cardiac catheterization (e.g., intracardiac thrombus).
* Impossibility of remote monitoring using an implantable Holter monitor or implantable defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mapping for the identification of stable reentrant domains with high activation frequency in persistent AF. | During procedure
  After performing cardiac CT, non-invasive mapping will be performed using ECGi non-invasive map system. The signals will be analyzed for real-time inverse solution calculations using: (i) the algorithms implemented in the commercial version of the equipment; and (ii) proprietary spectral fingerprint identification algorithms. In particular, non-invasive mapping will provide the fibrillation signal from both atria for the implementation of the calculations necessary for the spectral fingerprint study. The instantaneous phase will be computed by two methods: (i) by Hilbert transformation of the signal; and (ii) by phase calculation on the discrete frequencies identified in the power spectrogram.
  On the other hand, invasive mapping will be used to process bipolar and unipolar cardiac signals in order to analyze hierarchically organized patterns.
Effects of ablation of DFSAI > 0.8 domains on fibrillation dynamics and sustainability | During procedure
  * In patients in the active group, changes in fibrillation dynamics induced by CPVI and ablation of DFASI domains will be evaluated, as suggested by our preliminary results (Calvo D et al. Sci Rep. 2025 Dec 16;15(1):43892). Therefore, an experimental protocol will be carried out in which, after CPVI, each DFASI domain will be addressed sequentially. The following will be determined: a) changes in hierarchical organization levels, b) the formation of new DFASI domains; c) if AF ends after ablation, the termination mechanisms will be described. Once all ablation sets on the identified DFASI reentrant domains have been completed, noninvasive maps will be acquired under the effect of adenosine in order to compare fibrillatory dynamics under basal adenosine vs. post-ablation.
  * In patients in the control group, once CPVI is completed new noninvasive maps will be acquired to characterize basal and adenosine-induced fibrillatory dynamics.
Effects of ablation of reentrat domains of human ventricular fibrillation on arrhythmia inducibility. | Procedure
  Adapt the model to patients with ventricular arrhythmias such as polymorphic ventricular tachycardia and/or VF. After performing a cardiac CT scan, non-invasive mapping will be performed using ECGi non-invasive map system. The signals will be analyzed for real-time inverse solution calculations using: (i) the algorithms implemented in the commercial version of the equipment; and (ii) the algorithms for identifying reentrant domains and their correlation with hierarchical organization patterns. To this end, VF will be induced by programmed stimulation on two occasions in order to identify the hierarchical organization of the stability of rotational activity in terms of frequency. Ablation will follow and inducibility tested as measurement of efficacy.
Arrhythmia burden during Follow-up | 3, 6 and 12 months follow-up visits
  A subcutaneous Holter monitor will be implanted one month prior to the ablation procedure to mesure arrhythmia burden (Atrial fibrillation; number of recurrences and hours per day). Patients will be monitored continuously after the ablation procedure using remote subcutaneous Holter monitoring platforms and in person at cardiology consultations at 3, 6, and 12 months, at a minimum.
  Patients with VF ablation will be followed up after the ablation procedure on an ongoing basis using implantable defibrillator remote monitoring platforms and in person at cardiology consultations at least 3, 6, and 12 months after the procedure. The arrhythmia burden will be measure as a function of number of recurrences per follow-up time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided